CLINICAL TRIAL: NCT04039815
Title: Effects of Vitamin C, Thiamine and Hydrocortisone in Septic Shock: a Randomized, Controlled Trial
Brief Title: Vitamin C, Vitamin B1 and Steroid in Sepsis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 107133-F
Record Dates: First submitted 2018-12-11; First posted 2019-07-31 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2018-12

CONDITIONS: Sepsis, Severe
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: double blind, randomized-controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: as above
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABC group (Ascorbic acid-Vitamin B1-Hydrocortisone) group (Experimental): patients in study group, so called" ABC" (Ascorbic acid-Vitamin B1-Hydrocortisone) group, would receive intravenous Thiamine (200mg in 50 mL of 0.9% normal saline and was administered as a 30-min infusion every 12 hours for 4 days or until ICU discharge), Vitamin C (1.5g mixed in a 100-mL solution of normal saline and was administered as an infusion over 30 to 60 min every 6 hours for four days or until ICU discharge) as well as hydrocortisone 50mg every 6 hours (or other equivalent products) for 7 days
  Interventions: Drug: Ascorbic acid-Vitamin B1-Hydrocortisone
- normal saline group (Placebo Comparator): patients would receive 50mL 0.9% normal saline, 100 mL 0.9% normal saline with the same infusion rate and hydrocortisone dependent on the discretion of the attending physician
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ascorbic acid-Vitamin B1-Hydrocortisone — intravenous Thiamine (200mg in 50 mL of 0.9% normal saline and was administered as a 30-min infusion every 12 hours for 4 days or until ICU discharge), plus Vitamin C (1.5g mixed in a 100-mL solution of normal saline and was administered as an infusion over 30 to 60 min every 6 hours for four days or until ICU discharge) as well as hydrocortisone 50mg every 6 hours (or other equivalent products) for 7 days
  Arms: ABC group (Ascorbic acid-Vitamin B1-Hydrocortisone) group
Drug: Placebo — patients would receive 50mL 0.9% normal saline, 100 mL 0.9% normal saline with the same infusion rate and hydrocortisone dependent on the discretion of the attending physician
  Arms: normal saline group

SUMMARY:
A randomized controlled trial to test the synergic modulation effect of vitamin C, thiamine and hydrocortisone in patients with severe sepsis or septic shock.

DETAILED DESCRIPTION:
Management of sepsis bases on three components: infection control, haemodynamic stabilization and modulation of the septic response. Many clinical trials conducted agents to block the inflammatory cascade, such as corticosteroids, anti-endotoxins antibodies, tumor necrosis factor (TNF) antagonists, interleukin-1-receptor antagonists, and so on, but none has proven effective to date. A safe, effective, ready available therapy is desperately required. Thiamine is a key co-factor for pyruvate dehydrogenase, alpha-ketoglutarate dehydrogenase, and transketolase. All the three enzymes are required to complete Krebs Cycle to prevent from lactate production. Previous studies have found thiamine deficiency to be prevalent in septic shock and other critically ill conditions. One pilot study also proved patients with septic shock and baseline thiamine deficiency would have significant lower lactate level at 24 hours after administration of thiamine. HYPRESS (hydrocortisone for Prevention of Septic Shock) study failed to demonstrate an outcome benefit from a hydrocortisone infusion in patients with sepsis. Vitamin C is a potent antioxidant that directly scavenges oxygen free radicals, can restores other cellular antioxidants and plays a role in preserving endothelial function and microcirculatory flow as well. Though previous studies suggested that hydrocortisone and vitamin C alone have little impact on the clinical outcome of patients with sepsis. Vitamin C and hydrocortisone have many overlapping and synergic pathophysiologic effects in sepsis. Both drugs are required for the synthesis of catechlamines and increase vasopressor sensitivity. Both drugs can down-regulating the production of proinflammatory mediators, increase tight junctions between endothelial and epithelial cells, preserve endothelial function and microcirculatory flow. Marik et al published their study in CHEST (June 2017) resulting the benefits of combination of Vitamin B1, Vitamin C and hydrocortisone to severe sepsis and septic shock. However, small sample size and some bias due to imbalanced baseline and study method could confound the results. Herein, we would like to lead a randomized controlled trial to test the synergic modulation effect of vitamin C, thiamine and hydrocortisone in patients with severe sepsis or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* aged equal or over 20
* admitted to MICU due to severe sepsis or septic shock

Exclusion Criteria:

* Patients who are pregnant
* known history of Vitamin C , Vitamin B or hydrocortisone (or other equivalent products) allergy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint was the hospital survival. | 30 days
  hospital survival

SECONDARY OUTCOMES:
duration of vasopressor therapy | 72 hours
  duration of vasopressor therapy
requirement for renal replacement therapy in patients with acute kidney injury (AKI) | 72 hours
  requirement for renal replacement therapy in patients with acute kidney injury (AKI)
ICU length of stay (LOS) | 4 days
  ICU length of stay (days)
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  APACH II score (total 0~100) is a score to evaluate the mortality rate of ICU patients, higher values represent a worse outcome. It includes: (A) PaO2 (depending on FiO2) Temperature (rectal) Mean arterial pressure pH arterial Heart rate Respiratory rate Sodium (serum) Potassium (serum) Creatinine Hematocrit White blood cell count
  * (B) age points (score: 0~6)
  * (C) chronic health problems (liver cirrhosis, dialysis, COPD, congestive heart failure, immunocompromised)
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  PaO2 (depending on FiO2): mmHg
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  Temperature ( Celsius degrees)
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  Mean arterial pressure : mmHg
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  pH arterial
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  Heart rate: bpm
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  Respiratory rate: 1/min
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  Sodium (serum): mmol/L
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  Potassium (serum): mmol/L
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  Creatinine: mg/dL
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  Hematocrit: %
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  White blood cell count: 10 3/μL
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  age: years
change of Acute Physiology And Chronic Health Evaluation II (APACH II) score over the first 72 hours | 72 hours
  chronic health problems (liver cirrhosis, dialysis, COPD, congestive heart failure, immunocompromised): None: 0 point Non-surgical: 5 points Emergent operation: 5 points
Sequential Organ Failure Assessment score (SOFA score) over the first 72 hours | 72 hours
  PaO₂: mm Hg
Sequential Organ Failure Assessment score (SOFA score) over the first 72 hours | 72 hours
  Platelets: ×10³/µL
Sequential Organ Failure Assessment score (SOFA score) over the first 72 hours | 72 hours
  Glasgow Coma Scale: points 15: 0 13-14: +1 10-12: +2 6-9: +3 <6: +4
Sequential Organ Failure Assessment score (SOFA score) over the first 72 hours | 72 hours
  Bilirubin: mg/dL
Sequential Organ Failure Assessment score (SOFA score) over the first 72 hours | 72 hours
  Mean arterial pressure: mmHg
Sequential Organ Failure Assessment score (SOFA score) over the first 72 hours | 72 hours
  Creatinine: mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD are not to be shared with other researchers